CLINICAL TRIAL: NCT06729151
Title: Effect of Intradetrusor onabotulinumtoxinA Injection Versus Conservative Management on Female Sexual Function in Patients With Bladder Pain Syndrome
Status: Recruiting | Type: Observational
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: WRNMMC-2024-0450
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Bladder Pain Syndrome; Female Sexual Dysfunction
MeSH Terms: conditions — Cystitis, Interstitial | interventions — onabotulinum toxin A; Conservative Treatment; Diet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Controls: 49 healthy control patients complete the questionnaire packet once. No additional follow-up is completed.
- Bladder pain syndrome treated with conservative management: 55 patients with bladder pain syndrome who choose treatment with conservative management complete pre-treatment and 12-week post-treatment questionnaires.
  Interventions: Behavioral: Conservative management (dietary and behavioral)
- Bladder pain syndrome treated with bladder Botox: 55 patients with bladder pain syndrome who choose treatment with bladder Botox complete pre-treatment and 12-week post-treatment questionnaires.
  Interventions: Drug: Onabotulinum toxin A

INTERVENTIONS:
Drug: Onabotulinum toxin A — Cystoscopic injection of Onabotulinum toxin A per standard clinic protocol.
  Groups: Bladder pain syndrome treated with bladder Botox
Behavioral: Conservative management (dietary and behavioral) — Dietary and behavioral modifications consistent with recommendations from the American Urogynecological Society
  Groups: Bladder pain syndrome treated with conservative management

SUMMARY:
Interstitial cystitis/bladder pain syndrome (IC/BPS) is estimated to affect 3.3 to 7.9 million women aged 18 years and older in the United States. The American Urological Association (AUA) defines IC/BPS as "an unpleasant sensation (pain, pressure, discomfort) perceived to be related to the urinary bladder, associated with lower urinary tract symptoms of more than six weeks duration, in the absence of infection or other identifiable causes". IC/BPS significantly impacts quality of life, with the individual domains of sexual function, anxiety and depression, sleep quality and work productivity being specifically affected. Significant sexual dysfunction in women with IC/BPS has been consistently demonstrated across multiple international studies, with a prevalence ranging from 68% to 91%. In fact, among all patients with lower urinary tract symptoms, patients with a diagnosis of IC/BPS had the highest levels of impaired sexual function, mostly due to dyspareunia. Recommended treatments for IC/BPS include dietary and behavioral modifications, oral medications, bladder instillations, bladder hydrodistension, intradetrusor injection of onabotulinumtoxinA and major surgery. Scant research exists on how treating IC/BPS affects sexual function. We are conducting a prospective cohort study to assess for improvement in sexual function following intravesical onabotulinumtoxinA injection versus conservative management for IC/BPS.

The study will consist of three groups: intradetrusor onabotulinumtoxinA injection, conservative management and age-matched, healthy controls. All patients aged 18 years and older presenting to the Walter Reed National Military Medical Center (WRNMMC) Urogynecology clinic who are given a diagnosis of IC/BPS and have an O'Leary Sant index questionnaire scoring 13 or greater will be eligible for the study. The primary study outcome is change in the pre- and 12-week post-treatment Female Sexual Function Index (FSFI). The secondary outcomes will include changes in the pre- and post-treatment O'Leary Sant index, Patient Global Impression of Improvement (PGI-I), Patient Global Impression of Severity (PGI-S), Pelvic Organ Prolapse/Incontinence Sexual Questionnaire, IUGA-Revised (PISQ-IR), Visual analog pain scale and 24-hour bladder diary (number of daily voids, number of nightly voids, incontinence episode). Adverse events will be monitored, including urinary tract infection or need for urinary catheterization due to urinary retention within 12 weeks of start of treatment. The age-matched, healthy control group will complete only one set of questionnaires to serve as a baseline comparison to the IC/BPS groups. For between-groups comparisons, a sample size of 49 per group will have 80% power to detect a clinically important difference of 4 points if the standard deviation is 7 points, assuming a 5% two-sided significance level. We will therefore recruit 55 subjects per group to allow for approximately 10% attrition between the pre- and post-treatment assessments. This study will be powered to detect a difference between treatments groups, which has not yet been reported in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 years of age and older
* For bladder pain syndrome participants: O'Leary Sant score 13 or greater
* For healthy controls: O'Leary Sant score 12 or less
* DEERS eligible (care provided by military health care system)

Exclusion Criteria:

* Contraindications for bladder Botox
* Current use of alternative treatment for bladder pain syndrome
* Neurogenic bladder
* Other urinary tract disease
* Pelvic organ prolapse stage 3 or greater
* Pregnancy or breastfeeding
* Non-English speakers

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female-identifying individuals
Study Population: Patients with a clinical diagnosis of bladder pain syndrome and health controls without this diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function Index | Pre-treatment and 12 week post-treatment
  19-question survey encompassing several domains of sexual function in females

SECONDARY OUTCOMES:
O'Leary Sant Index | Pre-treatment and 12 week post-treatment
  Screening tool for bladder pain syndrome
Patient global impression of improvement (PGI-I) | 12 week post-treatment
Patient global impression of severity (PGI-S) | Pre-treatment and 12 week post-treatment
Pelvic pain and urgency/frequency symptom scale (PUF) | Pre-treatment and 12 week post-treatment
Female sexual distress scale-revised (FSDS-R) | Pre-treatment and 12 week post-treatment
Adverse events: UTI, urinary retention, additional treatment | 12 week post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States